CLINICAL TRIAL: NCT07375407
Title: The Effect of Aerobic Exercise and Physiological Ischemic Training on VEGF, Interleukin-6, Interleukin-10, Cardiorespiratory Fitness, Muscle Strength, and Quality of Life in Patients With Hypertension
Brief Title: Aerobic Exercise vs Physiological Ischemic Training in Stage 2 Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Arnengsih Nazir, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKFR-202502.02
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Hypertension, Grade 2
Keywords: Cardiorespiratory Fitness; Interleukin-6; Interleukin-10; Quality of Life; Vascular Endothelial Growth Factor A
MeSH Terms: conditions — Essential Hypertension; Lymphoma, Follicular | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (AE) (Experimental): Participants will perform a structured aerobic exercise program for 6 weeks, supervised by trained personnel. Outcomes measured include biomarkers (VEGF, IL-6, IL-10), cardiorespiratory fitness (VO2max, 6-minute walk distance), muscle strength (MVC), and quality of life (SF-36).
  Interventions: Behavioral: Aerobic Exercise (AE)
- Physiological Ischemic Training (PIT) (Experimental): articipants will perform a 6-week physiological ischemic training program, supervised by trained personnel. Outcomes measured include biomarkers (VEGF, IL-6, IL-10), cardiorespiratory fitness (VO2max, 6-minute walk distance), muscle strength (MVC), and quality of life (SF-36).
  Interventions: Behavioral: Physiological Ischemic Training (PIT)

INTERVENTIONS:
Behavioral: Aerobic Exercise (AE) — Participants will perform a structured aerobic exercise program for 6 weeks under supervision. The program is designed to improve cardiovascular fitness. Outcomes to be measured include biomarkers (VEGF, IL-6, IL-10), cardiorespiratory fitness (VO2max, 6-minute walk distance), muscle strength (MVC), and quality of life (SF-36)
  Arms: Aerobic Exercise (AE)
Behavioral: Physiological Ischemic Training (PIT) — Participants will perform a structured physiological ischemic training program for 6 weeks under supervision. The program is designed to modulate angiogenesis and inflammatory biomarkers. Outcomes to be measured include biomarkers (VEGF, IL-6, IL-10), cardiorespiratory fitness (VO2max, 6-minute walk distance), muscle strength (MVC), and quality of life (SF-36).
  Arms: Physiological Ischemic Training (PIT)

SUMMARY:
This study aims to compare the effects of aerobic exercise (AE) and physiological ischemic training (PIT) on inflammatory and angiogenesis biomarkers (VEGF, IL-6, IL-10), cardiorespiratory fitness, muscle strength, and quality of life in patients with grade 2 primary hypertension (HT2). This randomized controlled trial will involve 60 HT2 patients from Pratama and Utama Medika Antapani Clinic, who will be assigned to either AE or PIT groups. The intervention will last 6 weeks, and outcomes measured will include biomarker levels, VO2max, 6-minute walk distance (6-MWD), maximum voluntary contraction (MVC), and SF-36 questionnaire scores.

DETAILED DESCRIPTION:
Background: Grade 2 primary hypertension (HT2) can negatively affect cardiovascular health and quality of life. Physical exercise is a non-pharmacological intervention that may modulate inflammatory and angiogenesis biomarkers, as well as improve fitness and patient-reported outcomes. This study aims to compare the effects of aerobic exercise (AE) and physiological ischemic training (PIT) on HT2 patients.

Methods: This randomized controlled trial will include 60 HT2 patients from Pratama and Utama Medika Antapani Clinic. Participants will be randomly assigned to AE or PIT groups. The intervention will last 6 weeks. Outcomes to be measured include vascular endothelial growth factor (VEGF), interleukin-6 (IL-6), interleukin-10 (IL-10), cardiorespiratory fitness (VO2max, 6-minute walk distance [6-MWD]), muscle strength (maximum voluntary contraction [MVC]), and quality of life (SF-36 questionnaire).

ELIGIBILITY:
Inclusion Criteria:

1. Primary hypertension patients aged 18-65 years
2. Diagnosed with grade 2 primary hypertension
3. Willing to participate in the study

Exclusion Criteria:

1. Patients with unstable angina
2. Malignant arrhythmias and high atrioventricular block
3. Unstable hemodynamics
4. Uncontrolled hypertension
5. Acute pericarditis
6. Severe valvular heart disease
7. Chronic obstructive pulmonary disease
8. Cor pulmonale and pulmonary vascular disease
9. Thrombophlebitis
10. Intermittent claudication
11. Cognitive impairment
12. Uncooperative subjects
13. Subjects experiencing infection or inflammation
14. Subjects with neuromuscular disorders that may affect the study results
15. Subjects with musculoskeletal disorders that may affect the study results
16. Complications or comorbidities such as cerebrovascular disease, CAD, atheroma plaques on imaging, heart failure, PAD, and atrial fibrillation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Vascular Endothelial Growth Factor (VEGF) Level | Measured at baseline and after 6 weeks of intervention
  Change in circulating vascular endothelial growth factor (VEGF) concentration in peripheral blood, measured using a standardized laboratory assay, as an indicator of angiogenic response to the exercise intervention.

SECONDARY OUTCOMES:
Interleukin-6 (IL-6) Level | Baseline and 6 weeks
  Change in circulating interleukin-6 (IL-6) concentration in peripheral blood, measured using enzyme-linked immunosorbent assay (ELISA), as an indicator of systemic inflammatory response.
Interleukin-10 (IL-10) Level | Baseline and 6 weeks
  Change in circulating interleukin-10 (IL-10) concentration in peripheral blood, measured using enzyme-linked immunosorbent assay (ELISA), as an indicator of anti-inflammatory response.
6-Minute Walk Distance (6-MWD) | Baseline and 6 weeks
  Change in distance walked during the Six-Minute Walk Test (6MWT), measured in meters, as an assessment of functional exercise capacity. Higher distances indicate better functional capacity.
Muscle Strength (Maximum Voluntary Contraction, MVC) | Baseline and 6 weeks
  Change in maximal voluntary contraction (MVC), measured using a handheld or fixed dynamometer and expressed in Newtons (N) or kilograms (kg), as an indicator of muscular strength. Higher values indicate greater muscle strength.
Quality of Life (36-Item Short Form Health Survey, SF-36) | Baseline and 6 weeks
  Change in health-related quality of life assessed using the 36-Item Short Form Health Survey (SF-36). Scores for each domain range from 0 to 100, with higher scores indicating better perceived health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan sadikin general hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, after de-identification, will be made available to qualified researchers upon request. Requests will be reviewed by the study team and shared under data use agreements to ensure participant privacy and compliance with ethical guidelines.